CLINICAL TRIAL: NCT02119065
Title: PET/CT-Derived Hepatopulmonary Shunt Fraction Following Yttrium-90 Radioembolization
Brief Title: Pilot Study to Assess Lung Shunting of Yttrium-90 Microspheres Using PET/CT
Status: Active, not recruiting | Type: Observational
Sponsor: University of Cincinnati (Other)
Responsible Party: Principal Investigator, Michael V Knopp MD PhD, Principal Investigator, University of Cincinnati
Other Study IDs: OSU-13176; NCI-2014-00278 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2014-03-31; First posted 2014-04-21 (Estimated); Last update posted 2025-04-11 (Actual); Status verified 2025-04

CONDITIONS: Advanced Adult Primary Liver Cancer; Liver Metastases; Localized Unresectable Adult Primary Liver Cancer; Recurrent Adult Primary Liver Cancer
Keywords: Yttrium-90 Radioembolization; hepatic malignancy; hepatic metastatic disease
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Magnetic Resonance Spectroscopy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Health Services Research (PET/CT scan): Patients receive routine pre-therapy technetium Tc 99m-labeled macroaggregated albumin. Patients then undergo routine radioembolization with yttrium Y 90 resin microspheres. Within 36 hours after radioembolization, patients undergo PET/CT imaging.
  Interventions: Procedure: positron emission tomography; Procedure: computed tomography

INTERVENTIONS:
Procedure: positron emission tomography — Undergo PET/CT scan
  Other Names: PET; PET scan; tomography, positron emission
Procedure: computed tomography — Undergo PET/CT scan
  Other Names: tomography, computed

SUMMARY:
This pilot clinical trial studies positron emission tomography (PET)/computed tomography (CT) in finding beads after Yttrium-90 bead therapy in patients with primary liver cancer or cancer that has spread to the liver (metastatic) that can not be removed by surgery. Imaging procedures, such as PET/CT after Yttrium-90 bead therapy, may help see if the beads are present in the lung and compare the results with the pre-therapy imaging.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To estimate the absolute difference in post-therapy Yttrium-90 microsphere hepatopulmonary shunt fraction and the pre-therapy Technetium-99m macroaggregated albumin hepatopulmonary shunt fraction in patients with unresectable primary hepatic malignancy and hepatic metastatic disease.

SECONDARY OBJECTIVES:

I. To quantify and compare the pre-therapy Technetium-99m macroaggregated albumin particle sizes and post-therapy Yttrium-90 microsphere sizes.

OUTLINE:

Patients receive routine pre-therapy Technetium-99m macroaggregated albumin. Patients then undergo routine radioembolization with Yttrium-90 microspheres. Within 36 hours after radioembolization, patients undergo PET/CT imaging.

Available imaging, clinical, interventional and surgical follow-up data for 2 years after completion of enrollment in the study will be obtained.

ELIGIBILITY:
Inclusion Criteria:

* Patients who undergo intra-arterial hepatic 99mTc MAA evaluation in anticipation of 90Y microsphere radioembolization

Exclusion Criteria:

* Patients who are unable to give consent
* Prisoners

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The target population includes patients with unresectable liver metastases or malignancy who are referred to The Ohio State University Wexner Medical Center for Yttrium-90 microsphere radioembolization therapy.
Sampling Method: Non-Probability Sample
Enrollment: 6 (Actual)
Dates: Start 2014-01-30 (Actual); Primary Completion 2015-07-01 (Actual); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Absolute difference in post-therapy Yttrium-90 microsphere and pre-therapy Technetium-99m macroaggregated albumin hepatopulmonary shunt fraction values | Baseline to up to 36 hours after radioembolization
  Non-parametric Wilcoxon signed rank testing will be used to compare the 99mTc MAA and 90Y microsphere shunt fractions. Alternatively, a natural log transformation of the hepatopulmonary shunt fractions may be used to normalize these data for subsequent parametric paired t-test analysis.

SECONDARY OUTCOMES:
In vitro Technetium-99m macroaggregated albumin particle size and microsphere size for each patient | Baseline up to 24 months
  Descriptive statistical assessment of Technetium-99m macroaggregated albumin particle size and microsphere size for each patient (e.g., mean, median, standard deviation, distribution, etc.) will be performed.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Knopp, MD, PhD, Principal Investigator — Ohio State University Comprehensive Cancer Center
Locations (1):
- Arthur G. James Cancer Hospital and Solove Research Institute at Ohio State University Medical Center, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: The Jamesline — http://cancer.osu.edu